CLINICAL TRIAL: NCT04081571
Title: Prevalence of NAFLD and Correlation With Its Main Risk Factors Among Egyptian Multicenter National Study
Brief Title: Prevalence of NAFLD and Correlation With Its Main Risk Factors Among Egyptian
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Collaborators: Ain Shams University (Other); Mansoura University (Other); Alexandria University (Other); Fayoum University (Other); Tanta University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mona Hegazy, Professor of Internal Medicine Hepatology & gastroenterology Unit Faculty of medicine, Cairo University, Cairo University
Other Study IDs: 1001; N-41-2019 (Other: Cairo University ethical committee approval number)
Record Dates: First submitted 2019-07-30; First posted 2019-09-09 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: NAFLD; Insulin Resistance; Hepatic Steatosis
Keywords: NAFLD; Insulin Resistance; Hepatic Steatosis; EGYPTIAN
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Insulin Resistance; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Getting a rough indicator about the prevalence of different grade of severity of NAFLD (NASH & liver fibrosis), and Correlate the severity of fatty liver with different serological risk factors of metabolic syndrome and diseases progression as well as the prevalence of hepatocellular carcinoma related to NAFLD with the use of ; nutritional assessment designed and conducted by the investigators in this research, simple blood test (lipid profile and blood sugar), and easy cheap non-invasive radiological tool as screening to predict NASH.

DETAILED DESCRIPTION:
This study is a prospective cross-sectional Multicenter National study, will include 1080 participants with BMI ≥ 24kg/m 2 with or without elevated liver enzymes. All will be subjected to; dietary history by already prepared food quality and quantity questionnaire, anthropometric data (BMI & waist circumference), Clinical examination, Laboratory work include: total lipid profile (LDL-C, HDL-C, VLDL (very low-density lipoprotein)& TGs (Triglyceride)), fasting blood glucose and insulin (HOMA-IR (Insulin Resistance) will be calculated), HbA1c%, liver biochemistry tests (ALT, GGT (Gammaglutamyl transpeptidase), AST (aspartate aminotransferase), and bilirubin), Liver function testes (INR & albumin), HCV (Hepatitis C virus) antibody, HBV (Hepatitis B virus) surface antigen, TSH (thyroid-stimulating hormone) , Free T3 & T4 will be done for all participants. Imaging; Liver ultrasound including measurement of the subcutaneous fat in front of the left lobe of liver as well as at the umbilical region and assessment of liver stiffness by Fibroscan.

The novelty of this study is that, if it showed a successful outcome, the investigators will get a rough indicator about the prevalence of different grade of severity of NAFLD, and Correlate the severity of fatty liver with different risk factors of metabolic syndrome and life style modifications among Egyptians, and trying to confirm the great variability between different races regarding BMI classes and overweight & obesity cut-off values, confirming the high level of insulin resistance in non-diabetic participants with NAFLD compared to other races, identify types of food that are at risk for development and progression of NAFLD thus getting a healthy food recommendations for Egyptians and get a recommendation for another studies for metabolic syndrome redefinition with NAFLD part of it (not just considering as known in the present time), and working on the Triglycerides, LDL, and HDL cut off values. investigators also hope through this research to modify dietary habits in the Egyptian society encouraging healthy nutrition through dietary assessment (already prepared food quality and quantity questionnaire), that can lead to not only NAFLD but also progress to NASH, so participants can promote healthy dietary habits and proper life style among different health care providers thus decreasing incidence of obesity, one of main risk factors of fatty liver diseases and its consequences especially Hepatocellular Cancer.

Investigators also hope through this research to modify dietary habits in the Egyptian society encouraging healthy nutrition through promoting professional nutritional assessment and questionnaire among different health care providers thus decreasing incidence of obesity, one of main risk factors of fatty liver diseases and its consequences especially Hepatocellular Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants with following criteria: age: 18-60 years and both sexes
* Any participant with BMI more than or equal to 24kg/m2 (overweight and obese according to Chinese cut off values)

Exclusion Criteria:

* Any hepatic diseases including e.g. Hepatitis C, Hepatitis B, autoimmune hepatitis
* Pregnant females
* Alcohol intake
* Antibiotic use within the previous 3 months
* Patients had acute or chronic health diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study is a prospective cross-sectional Multicenter National study, including 1080 participants with BMI ≥ 24kg/m diagnosed with a high probability of NAFLD using ultrasound with or without elevated liver enzymes
Sampling Method: Probability Sample
Enrollment: 1080 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of different grads of severity of NAFLD and Correlation with Its main risk Factors among Egyptians | April 2019 to March 2021
  In the Middle East, till the present time, no data about the incidence, prevalence of NAFLD early identification of patients with NASH prior to the onset of advanced fibrosis would be helpful in guiding aggressive interaction.
Dietary history | April 2019 to March 2021
  Food Frequency Checklist will be done. Mean daily consumption of selected food items will be calculated
  Optimal level of intake and optimal range of intake :
  1. Fruits: 250 g (200-300) per day
  2. Vegetables:360 g (290-430) per day
  3. Grains:125 g (100-150) per day
  4. Legumes : 60 g (50-70) per day
  5. Milk & milk products: 435 g (350-520) per day
  6. Sodium: 3 g (1-5) per day
  7. Sugar & sweetened products:3 g (0-5) per day
  8. Meats : 23 g (18-27) per day)
  9. Processed meat:2 g (0-4) per day
  10. Sea foods & omega 3 fatty acids : 250 mg (200-300) per day
  11. Nuts &seeds :21 g (16-25) per day
  12. Polyunsaturated oils :11% (9-13) of total daily energy
  13. Trans fat-margarine :0·5% (0·0-1·0) of total daily energy
  14. Dietary fibers :24 g (19-28) per day
  15. Calcium :1,25 g(1,00-1.5g) per day
Risk factors of NAFLD | April 2019 to March 2021
  The prevalence of NAFLD has risen rapidly in parallel with the dramatic rise in population levels of obesity and diabetes and the entire world follow the European BMI classification and the parameters for metabolic syndrome diagnosis, except for the modification done by china.

SECONDARY OUTCOMES:
Prevalence of NAFLD among different ethnic groups | April 2019 to March 2020
  Trying to confirm the great variability between different races regarding BMI classes and overweight & obesity cut-off values
Prevalence of Insulin resistance | April 2019 to March 2020
  Confirming the high level of insulin resistance in non-diabetic compared to other races
Prevalence of Metabolic syndrome | April 2019 to March 2020
  if all the patients diagnosed as have metabolic syndrome according to international criteria, have NAFLD. Also the results of the present study will cover the cut of value of waist circumference in criteria of metabolic syndrome and the present study will show that those cut-of applied on Egyptians or not. So a recommendation for another studies for metabolic syndrome redefinition with NAFLD part of it (not just considering as known in the present time), and working on the Triglycerides, HDL cut off values & changing blood sugar with the HOMA-IR (Homeostatic model assessment-insulin resistance) in Egyptians will be one of the present study expected outcomes recommendation
NASH staging | April 2019 to March 2020
  Trying to get a cut-off value for LSFT (subcutaneous fat in front of left lobe of liver) and USFT (subcutaneous fat at umbilical region) as the investigators previous published work concluded that: LSFT, and USFT had high sensitivity and specificity as simple non-invasive screening method to identify the presence of NASH as prediction of NAFLD progression, so working on a large scale study as a novel method for easy identification and staging of NAFLD.

CONTACTS AND LOCATIONS:
Overall Officials: Mona A Hegazy, MD, Principal Investigator — Professor of Internal Medicine Hepatology, Faculty of medicine, Cairo University; Ahmed M Abdul Ghani, MD, Study Director — Lecturer of Internal Medicine & Hepatology, Faculty of Medicine, Cairo University
Locations (1):
- Faculty of Medicine Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Vuppalanchi R, Chalasani N. Nonalcoholic fatty liver disease and nonalcoholic steatohepatitis: Selected practical issues in their evaluation and management. Hepatology. 2009 Jan;49(1):306-17. doi: 10.1002/hep.22603. PMID 19065650
- [Background] de Alwis NM, Day CP. Non-alcoholic fatty liver disease: the mist gradually clears. J Hepatol. 2008;48 Suppl 1:S104-12. doi: 10.1016/j.jhep.2008.01.009. Epub 2008 Feb 4. PMID 18304679
- [Background] Marchesini G, Moscatiello S, Agostini F, Villanova N, Festi D. Treatment of non-alcoholic fatty liver disease with focus on emerging drugs. Expert Opin Emerg Drugs. 2011 Mar;16(1):121-36. doi: 10.1517/14728214.2011.531700. PMID 21352073
- [Background] Loomba R, Sanyal AJ. The global NAFLD epidemic. Nat Rev Gastroenterol Hepatol. 2013 Nov;10(11):686-90. doi: 10.1038/nrgastro.2013.171. Epub 2013 Sep 17. PMID 24042449
- [Background] Smith BW, Adams LA. Non-alcoholic fatty liver disease. Crit Rev Clin Lab Sci. 2011 May-Jun;48(3):97-113. doi: 10.3109/10408363.2011.596521. PMID 21875310
- [Background] Zhan Y, Zhao F, Xie P, Zhong L, Li D, Gai Q, Li L, Wei H, Zhang L, An W. Mechanism of the effect of glycosyltransferase GLT8D2 on fatty liver. Lipids Health Dis. 2015 May 8;14:43. doi: 10.1186/s12944-015-0040-3. PMID 25952508
- [Background] White DL, Kanwal F, El-Serag HB. Association between nonalcoholic fatty liver disease and risk for hepatocellular cancer, based on systematic review. Clin Gastroenterol Hepatol. 2012 Dec;10(12):1342-1359.e2. doi: 10.1016/j.cgh.2012.10.001. Epub 2012 Oct 4. PMID 23041539
- [Background] Lazo M, Clark JM. The epidemiology of nonalcoholic fatty liver disease: a global perspective. Semin Liver Dis. 2008 Nov;28(4):339-50. doi: 10.1055/s-0028-1091978. Epub 2008 Oct 27. PMID 18956290
- [Background] Zhou B; Coorperative Meta-Analysis Group Of Working Group On Obesity In China. [Prospective study for cut-off points of body mass index in Chinese adults]. Zhonghua Liu Xing Bing Xue Za Zhi. 2002 Dec;23(6):431-4. Chinese. PMID 12667353
- [Background] Omagari K, Kadokawa Y, Masuda J, Egawa I, Sawa T, Hazama H, Ohba K, Isomoto H, Mizuta Y, Hayashida K, Murase K, Kadota T, Murata I, Kohno S. Fatty liver in non-alcoholic non-overweight Japanese adults: incidence and clinical characteristics. J Gastroenterol Hepatol. 2002 Oct;17(10):1098-105. doi: 10.1046/j.1440-1746.2002.02846.x. PMID 12201871
- [Background] Fan JG, Farrell GC. Epidemiology of non-alcoholic fatty liver disease in China. J Hepatol. 2009 Jan;50(1):204-10. doi: 10.1016/j.jhep.2008.10.010. Epub 2008 Nov 6. PMID 19014878
- [Background] Lee JY, Kim KM, Lee SG, Yu E, Lim YS, Lee HC, Chung YH, Lee YS, Suh DJ. Prevalence and risk factors of non-alcoholic fatty liver disease in potential living liver donors in Korea: a review of 589 consecutive liver biopsies in a single center. J Hepatol. 2007 Aug;47(2):239-44. doi: 10.1016/j.jhep.2007.02.007. Epub 2007 Mar 6. PMID 17400323
- [Background] Heron M. Deaths: Leading Causes for 2014. Natl Vital Stat Rep. 2016 Jun;65(5):1-96. PMID 27376998
- [Background] Guerrero R, Vega GL, Grundy SM, Browning JD. Ethnic differences in hepatic steatosis: an insulin resistance paradox? Hepatology. 2009 Mar;49(3):791-801. doi: 10.1002/hep.22726. PMID 19105205
- [Background] Pan JJ, Fallon MB. Gender and racial differences in nonalcoholic fatty liver disease. World J Hepatol. 2014 May 27;6(5):274-83. doi: 10.4254/wjh.v6.i5.274. PMID 24868321
- [Background] Assy N, Kaita K, Mymin D, Levy C, Rosser B, Minuk G. Fatty infiltration of liver in hyperlipidemic patients. Dig Dis Sci. 2000 Oct;45(10):1929-34. doi: 10.1023/a:1005661516165. PMID 11117562
- [Background] Schwimmer JB, Deutsch R, Rauch JB, Behling C, Newbury R, Lavine JE. Obesity, insulin resistance, and other clinicopathological correlates of pediatric nonalcoholic fatty liver disease. J Pediatr. 2003 Oct;143(4):500-5. doi: 10.1067/S0022-3476(03)00325-1. PMID 14571229
- [Background] Salman A, Hegazy M, AbdElfadl S. Combined Adiponectin Deficiency and Resistance in Obese Patients: Can It Solve Part of the Puzzle in Nonalcoholic Steatohepatitis. Open Access Maced J Med Sci. 2015 Jun 15;3(2):298-302. doi: 10.3889/oamjms.2015.057. Epub 2015 May 30. PMID 27275239
- [Background] Hegazy M, Abo-Elfadl S, Mostafa A, Ibrahim M, Rashed L, Salman A. Serum Resistin Level and Its Receptor Gene Expression in Liver Biopsy as Predictors for the Severity of Nonalcoholic Fatty Liver Disease. Euroasian J Hepatogastroenterol. 2014 Jul-Dec;4(2):59-62. doi: 10.5005/jp-journals-10018-1102i. Epub 2014 Jul 28. PMID 29699348
- [Background] Hegazy MA, Samy MA, Tawfik A, Naguib MM, Ezzat A, Behiry ME. Abdominal subcutaneous fat thickness and homeostasis model assessment of insulin resistance as simple predictors of nonalcoholic steatohepatitis. Diabetes Metab Syndr Obes. 2019 Jul 11;12:1105-1111. doi: 10.2147/DMSO.S202343. eCollection 2019. PMID 31372020